CLINICAL TRIAL: NCT05470101
Title: An Open-label, Positron Emission Tomography (PET) Study to Evaluate Brain Receptor Occupancy, Safety, Tolerability, and Pharmacokinetics After Single Oral Doses of ITI-333 in Healthy Subjects
Brief Title: A PET Study Following a Single Oral Dose of ITI-333 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: ITI-333-003
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1: ITI-333 2.25 mg (Experimental)
  Interventions: Drug: ITI-333
- Cohort A2: ITI-333 dose to be determined based on Cohort A1 (Experimental)
  Interventions: Drug: ITI-333
- Cohort A3: ITI-333 dose to be determined based on Cohort A1 and A2 (Experimental)
  Interventions: Drug: ITI-333
- Cohort A4: ITI-333 dose to be determined based on Cohort A1, A2 and A3 (Experimental)
  Interventions: Drug: ITI-333

INTERVENTIONS:
Drug: ITI-333 — ITI-333 oral solution

SUMMARY:
This is an open-label, single-dose study of up to 4 dose levels of ITI-333 in healthy male and female subjects. Each cohort will enroll 6 subjects. Subjects will have a baseline PET/CT scan and a postdose PET/CT scan using [14C]-MDL100907 to characterize 5-HT2A receptor occupancy

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 and 45 years old (inclusive);
* BMI inclusive of 18.0-32.0 kg/m2 at screening and a minimum weight of 50 kg;
* Willing to be confined to the clinical research unit for the duration of the inpatient period of the study;

Exclusion Criteria:

* Clinically significant abnormality within 2 years of Screening that in the Investigator's opinion may place the subject at risk or interfere with study outcome variables; this includes, but is not limited to, history of or current cardiac, hepatic, renal, neurologic, gastrointestinal (including history of gastric bypass), pulmonary, endocrinologic, hematologic, or immunologic disease or history of malignancy;
* Clinically significant abnormal findings in vital sign assessments, including blood oxygen saturation (SpO2) < 96% and respiratory rate < 12 breaths per min;
* History of psychiatric condition that in the Investigator's opinion may be detrimental to participation in the study;
* Any condition which would preclude MRI or PET/CT examination (eg, implanted metal, claustrophobia, unable to fit in PET/CT or MRI scanners).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: 5-HT2A receptor occupancy (RO) using [11C]-MDL100907 | baseline 90-minute PET scan between Day -10 and Day -1, and a 90-minute PET scan starting at approximately 1 hour postdose
Pharmacokinetics: AUC0-t | predose and multiple timepoints up to 24 hours postdose
  Area under the plasma concentration time curve from time zero to the last measurable of concentration of ITI-333
Pharmacokinetics: Cmax | predose and multiple timepoints up to 24 hours postdose
  Maximum observed plasma concentration
Pharmacokinetics: Tmax | predose and multiple timepoints up to 24 hours postdose
  Time to reach maximum observed plasma concentration

SECONDARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events | up to 30 days after last dose
Change from baseline in systolic and diastolic blood pressure | Up to Day 7
Change from baseline in ECG QT interval | Up to Day 7
Change from baseline in aspartate aminotransferase | Up to Day 7
Change from baseline in alanine aminotransferase | Up to Day 7

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Site 2, Creve Coeur, Missouri
  - Clinical Site 1, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No